CLINICAL TRIAL: NCT05569044
Title: Effects of Oral Rehydration Solutions in Healthy Adult Athletes
Brief Title: Oral Rehydration Solutions in Healthy Adult Athletes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment Challenges
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BL67
Record Dates: First submitted 2022-09-19; First posted 2022-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hydration
MeSH Terms: interventions — Control Groups; World Health Organization oral rehydration solution; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): No intervention
  Interventions: Other: Control Group
- Oral Rehydration Solution (Experimental): ORS with carbohydrate
  Interventions: Other: Oral Rehydration Solution
- Water (Experimental): Water with flavor
  Interventions: Other: Water

INTERVENTIONS:
Other: Control Group — No intervention
  Arms: Control Group
Other: Oral Rehydration Solution — Participants will be administered ORS during one of the study visits
  Arms: Oral Rehydration Solution
Other: Water — Participants will be administered water during one of the study visits
  Arms: Water

SUMMARY:
This is a prospective, randomized, controlled, crossover study to determine the benefits of adult athletes consuming an oral rehydration solution (ORS) with exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years of age.
* Body fat percentage ≤17% for males and ≤24% for females.
* Male or non-pregnant, non-lactating female, at least 6 months postpartum prior to screening visit.
* Cycling VO2max in range of 45-53 mL O2/kg/min for males or 36-43 mL O2/kg/min for females.
* If female, participant has a regular menstrual cycle, >21 days and <35 days in length.
* Willing to consume grape-flavored beverages during the study.
* If on chronic medication such as lipid-lowering, thyroid medication or hormone therapy, the dosage must be constant for at least 2 months prior to screening and baseline visit.
* Weight-stable for the two months prior to screening visit
* Voluntarily signed and dated an informed consent form (ICF), approved by an IRB, and provided Health Insurance Portability and Accountability Act (HIPAA) or other applicable privacy regulation authorization prior to any participation in the study.
* No known intolerance or allergy to ingredients in study products.
* Willing to refrain from using saunas or hot tubs for the duration of the study.
* Willing to follow study procedures and complete any forms or assessments needed during the study.

Exclusion Criteria:

* Athlete in a weight-conscious sport such as but not limited to wrestling, powerlifting, boxing, rowing, gymnastics or any martial arts.
* Currently, and for the past 4 weeks or longer: running >40 miles per week on average, cycling >80 miles per week on average or swimming >20,000 yards per week on average.
* Participating in another study that has not been approved as a concomitant study.
* Uses any form of tobacco or nicotine, or other controlled substance not prescribed by a physician.
* Previous history with heat illness or injury that resulted in a visit to a medical center.
* Experienced a serious musculoskeletal injury or surgery in the past 6 months that poses a risk during the trial, according to the study investigator.
* Eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures.
* Currently taking or has taken antibiotics within 6 weeks of enrollment.
* Currently taking or has taken a diuretic within 1 week of enrollment.
* Diagnosed with the following according to medical records, self-report or according to the clinician's judgment:

  * Acute or chronic infections including but not restricted to respiratory infections, diarrhea, Hepatitis B or C, HIV infection or tuberculosis
  * Severe gastrointestinal disorders such as celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis
  * Cardiovascular, metabolic [including diabetes], renal, hepatic, or respiratory disease
  * Active malignancy
  * Polycystic ovary disease
* Any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Anaerobic Power | Through Study completion, an average of 6 weeks
  Change in cycling power

SECONDARY OUTCOMES:
Body Mass | Through Study completion, an average of 6 weeks
  Body mass loss
Power Output | Through Study completion, an average of 6 weeks
  Mean cycling power
Rating of Perceived Exertion (RPE) | Through Study completion, an average of 6 weeks
  Participant completed scale of perceived exertion from 6 (no exertion at all) to 20 (maximum exertion)
Leg Strength | Through Study completion, an average of 6 weeks
  Measured by dynamometer
Muscular Force | Through Study completion, an average of 6 weeks
  Change in isometric muscular contractions

OTHER OUTCOMES:
Reaction Time | Through Study completion, an average of 6 weeks
  Change in reaction time
Muscular Endurance | Through Study completion, an average of 6 weeks
  Measured by dynamometer
Muscular Strength | Through Study completion, an average of 6 weeks
  Change in hand grip strength
Hydration Status Plasma | Through Study completion, an average of 6 weeks
  Change in plasma osmolality
Hydration Status Urine | Through Study completion, an average of 6 weeks
  Change in urine osmolality
Hydration Status Saliva | Through Study completion, an average of 6 weeks
  Change in saliva osmolality
Blood Biomarkers Creatinine | Through Study completion, an average of 6 weeks
  Change in concentrations of creatinine
Blood Biomarkers Cytokines | Through Study completion, an average of 6 weeks
  Change in concentrations of cytokines
Blood Biomarkers Glucose | Through Study completion, an average of 6 weeks
  Change in concentrations of glucose
Blood Biomarkers Insulin | Through Study completion, an average of 6 weeks
  Change in concentrations of insulin
Body Temperature | Through Study completion, an average of 6 weeks
  Change in degrees Celsius
Heart Rate | Through Study completion, an average of 6 weeks
  Change in heart rate
Profile of Mood States | Through Study completion, an average of 6 weeks
  Participant completed questionnaire of 35 feelings rated from 0 (not at all) to 4 (extremely)
Thirst Sensation Scale | Through Study completion, an average of 6 weeks
  Participant completed thirst question related from 1 (not thirsty at all) to 7 (very, very thirsty)
Gagge Thermal Scale | Through Study completion, an average of 6 weeks
  Change in participant reported comfort (scored 1 Comfortable to 4 Very Uncomfortable) and sensation (scored 1 Cold to 7 Hot)
Palatability | Through Study completion, an average of 6 weeks
  3 participant completed Likert scale questions scored from 1 (Dislike/Not at all) to 9 (Extremely)
Adverse Events | Through Study completion, an average of 6 weeks
  Participant experienced adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, MPH, Study Chair — Abbott Nutrition
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No